CLINICAL TRIAL: NCT03827798
Title: A Randomized, Subject and Investigator Blinded, Placebo-controlled and Multi-center Platform Study, to Assess Efficacy and Safety of Different Investigational Drugs in Patients With Moderate to Severe Hidradenitis Suppurativa
Brief Title: Study of Efficacy and Safety of Investigational Treatments in Patients With Moderate to Severe Hidradenitis Suppurativa
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCFZ533H12201BC
Record Dates: First submitted 2019-01-31; First posted 2019-02-01 (Actual); Results first posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Hidradenitis Suppurativa
Keywords: Hidradenitis suppurativa; acne inversa; platform study
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — iscalimab; remibrutinib; ianalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Cohort A - CFZ533 600 mg (Experimental): CFZ533 600 mg administered subcutaneous (s.c) weekly for 4 weeks, followed by bi-weekly until Week 15.
  Interventions: Drug: CFZ533
- Cohort B - LYS006 20 mg (Experimental): LYS006 20 mg administered orally twice per day until Week 16.
  Interventions: Drug: LYS006
- Cohort A - Placebo to CFZ533 (Placebo Comparator): Placebo administered subcutaneous (s.c) weekly for 4 weeks, followed by bi-weekly until Week 15.
  Interventions: Drug: Placebo to CFZ533
- Cohort B - Placebo to LYS006 (Placebo Comparator): Placebo administered orally twice per day until Week 16.
  Interventions: Drug: Placebo to LYS006
- Cohort C - MAS825 300 mg (Experimental): MAS825 300 mg administered s.c. bi-weekly for 4 weeks, followed by monthly until Week 13.
  Interventions: Drug: MAS825
- Cohort C - Placebo to MAS825 (Placebo Comparator): Placebo administered s.c. bi-weekly for 4 weeks, followed by monthly until Week 13.
  Interventions: Drug: Placebo to MAS825
- Cohort D - LOU064 25mg (Experimental): LOU064 25 mg administered orally twice per day until Week 16.
  Interventions: Drug: LOU064 25mg
- Cohort D - LOU064 100mg (Experimental): LOU064 100 mg administered orally twice per day until Week 16.
  Interventions: Drug: LOU064 100mg
- Cohort D - Placebo to LOU064 (Placebo Comparator): Placebo administered orally twice per day until Week 16.
  Interventions: Drug: Placebo to LOU064
- Cohort E - VAY736 300 mg (Experimental): VAY736 300 mg administered s.c every 4 weeks until Week 13.
  Interventions: Drug: VAY736
- Cohort E - Placebo to VAY736 (Placebo Comparator): Placebo administered s.c every 4 weeks until Week 13.
  Interventions: Drug: Placebo to VAY736

INTERVENTIONS:
Drug: CFZ533 — CFZ533 600 mg administered subcutaneous (s.c) weekly for 4 weeks, followed by bi-weekly until Week 15.
  Other Names: iscalimab
  Arms: Cohort A - CFZ533 600 mg
Drug: Placebo to CFZ533 — Placebo administered subcutaneous (s.c) weekly for 4 weeks, followed by bi-weekly until Week 15.
  Arms: Cohort A - Placebo to CFZ533
Drug: LYS006 — LYS006 20 mg administered orally twice per day until Week 16.
  Arms: Cohort B - LYS006 20 mg
Drug: Placebo to LYS006 — Placebo administered orally twice per day until Week 16.
  Arms: Cohort B - Placebo to LYS006
Drug: MAS825 — MAS825 300 mg administered s.c. bi-weekly for 4 weeks, followed by monthly until Week 13.
  Arms: Cohort C - MAS825 300 mg
Drug: Placebo to MAS825 — Placebo administered s.c. bi-weekly for 4 weeks, followed by monthly until Week 13.
  Arms: Cohort C - Placebo to MAS825
Drug: LOU064 25mg — LOU064 25 mg administered orally twice per day until Week 16.
  Other Names: remibrutinib
  Arms: Cohort D - LOU064 25mg
Drug: LOU064 100mg — LOU064 100 mg administered orally twice per day until Week 16.
  Other Names: remibrutinib
  Arms: Cohort D - LOU064 100mg
Drug: Placebo to LOU064 — Placebo administered orally twice per day until Week 16.
  Arms: Cohort D - Placebo to LOU064
Drug: VAY736 — VAY736 300 mg administered s.c every 4 weeks until Week 13.
  Other Names: ianalumab
  Arms: Cohort E - VAY736 300 mg
Drug: Placebo to VAY736 — Placebo administered s.c every 4 weeks until Week 13.
  Arms: Cohort E - Placebo to VAY736

SUMMARY:
The main purpose of this study is to assess preliminary efficacy and safety of CFZ533/iscalimab (Cohort A), LYS006 (Cohort B), MAS825 (Cohort C), LOU064/remibrutinib (Cohort D) and VAY736/ianalumab (Cohort E) in patients with moderate to severe hidradenitis suppurativa and to determine if CFZ533, LYS006, MAS825, LOU064 and VAY736 have an adequate clinical profile for further clinical development.

DETAILED DESCRIPTION:
This is a randomized, subject and investigator-blinded, placebo-controlled, multi-center and parallel-group non-confirmatory study to assess the efficacy, safety and tolerability of five investigational drugs, CFZ533 (iscalimab), LYS006, MAS825, LOU064 (remibrutinib) and VAY736 (ianalumab) in subjects with moderate to severe hidradenitis suppurativa.

All participants from Cohorts A, B and C had planned a 16-week treatment period and 12-week safety follow up period. All participants for Cohort D had planned a 16-week treatment period and 4-week safety follow up period.

All participants for Cohort E had planned a 16-week treatment period and a mandatory 16-week safety follow-up period, plus a conditional follow-up period for up to 84 weeks for a total maximum follow up period of 2 years. Cohorts A-D are completed and Cohort E is ongoing.

ELIGIBILITY:
Inclusion Criteria:

* Patients with moderate to severe HS based on the number of lesions, fistulae and anatomical areas involved
* Minimal body weight of 50 kg
* Able to communicate well with the investigator and understand and comply with the requirements of the study, and the ability and willingness to conduct study visits as per the study schedule

Exclusion Criteria:

* Use of other investigational drugs at the time of screening or before
* Women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception
* Pregnant or lactating women

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2024-12-04 (Actual); Study Completion 2026-12-11 (Estimated)

CONTACTS AND LOCATIONS:
Locations (36):
- United States (8):
  - Olympian Clinical Research, Clearwater, Florida
  - Park Avenue Dermatology PA, Orange Park, Florida
  - University Of South Florida, Tampa, Florida
  - Advanced Medical Research, Sandy Springs, Georgia
  - NorthShore University Health System, Evanston, Illinois
  - Dawes Fretzin Clinical Rea Group, Indianapolis, Indiana
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Medical University of South Carolina MUSC, Charleston, South Carolina
- Novartis Investigative Site, Graz, Austria
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Prague, Prague 1, Czechia
- Denmark (2):
  - Novartis Investigative Site, Copenhagen
  - Novartis Investigative Site, Roskilde
- France (6):
  - Novartis Investigative Site, Antony
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rouen
- Germany (4):
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Schwerin
- Hungary (4):
  - Novartis Investigative Site, Pécs, Baranya
  - Novartis Investigative Site, Debrecen, Hajdu Bihar Megye
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Szeged
- Novartis Investigative Site, Kopavogur, Iceland
- Netherlands (2):
  - Novartis Investigative Site, Rotterdam, South Holland
  - Novartis Investigative Site, Groningen
- Spain (6):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Sabadell, Barcelona
  - Novartis Investigative Site, Manises, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Las Palmas GC
  - Novartis Investigative Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in 36 investigative sites in 11 countries.
Pre-assignment Details: The study consisted of a screening period of up to 35 days. After last dose of study treatment patients could enter the post-treatment follow-up.
Groups:
- Cohort D - LOU064 25 mg: LOU064 25 mg administered orally twice per day until Week 16.
- Cohort D - LOU064 100 mg: LOU064 100 mg administered orally twice per day until Week 16.
Period: Treatment Epoch
Arm/Group | Cohort A - CFZ533 600 mg | Cohort A - Placebo to CFZ533 | Cohort B - LYS006 20 mg | Cohort B - Placebo to LYS006 | Cohort C - MAS825 300 mg | Cohort C - Placebo to MAS825 | Cohort D - LOU064 25 mg | Cohort D - LOU064 100 mg | Cohort D - Placebo to LOU064 | Cohort E - VAY736 300 mg | Cohort E - Placebo to VAY736
Started | 29 | 16 | 27 | 13 | 33 | 10 | 33 | 33 | 11 | 32 | 11
Completed | 25 | 12 | 20 | 9 | 29 | 9 | 29 | 26 | 8 | 23 | 10
Not Completed | 4 | 4 | 7 | 4 | 4 | 1 | 4 | 7 | 3 | 9 | 1
Not completed — Adverse Event | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 3 | 4 | 1 | 2 | 1 | 4 | 3 | 2 | 8 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Period: Entered Post-treatment Follow-up
Arm/Group | Cohort A - CFZ533 600 mg | Cohort A - Placebo to CFZ533 | Cohort B - LYS006 20 mg | Cohort B - Placebo to LYS006 | Cohort C - MAS825 300 mg | Cohort C - Placebo to MAS825 | Cohort D - LOU064 25 mg | Cohort D - LOU064 100 mg | Cohort D - Placebo to LOU064 | Cohort E - VAY736 300 mg | Cohort E - Placebo to VAY736
Started | 26 | 12 | 21 | 9 | 28 | 9 | 30 | 27 | 8 | 23 | 10
Completed | 24 | 11 | 19 | 8 | 26 | 7 | 30 | 25 | 8 | 0 | 1
Not Completed | 2 | 1 | 2 | 1 | 2 | 2 | 0 | 2 | 0 | 23 | 9
Not completed — Follow up ongoing | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 21 | 9
Not completed — Lost to Follow-up | 1 | 0 | 1 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A - CFZ533 600 mg | Cohort A - Placebo to CFZ533 | Cohort B - LYS006 20 mg | Cohort B - Placebo to LYS006 | Cohort C - MAS825 300 mg | Cohort C - Placebo to MAS825 | Cohort D - LOU064 25 mg | Cohort D - LOU064 100 mg | Cohort D - Placebo to LOU064 | Cohort E - VAY736 300 mg | Cohort E - Placebo to VAY736 | Total
Number analyzed (Participants) | 29 | 16 | 27 | 13 | 33 | 10 | 33 | 33 | 11 | 32 | 11 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (8.68) | 41.4 (9.54) | 36.4 (9.62) | 36.5 (13.29) | 39.5 (8.22) | 36.9 (10.26) | 35.6 (10.84) | 35.3 (10.99) | 44.1 (7.83) | 34.6 (8.35) | 33.1 (11.26) | 37.0 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 10 | 17 | 7 | 19 | 3 | 18 | 20 | 3 | 17 | 4 | 134
  Male | 13 | 6 | 10 | 6 | 14 | 7 | 15 | 13 | 8 | 15 | 7 | 114
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian: Asian | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 4
  Asian: Black Or African American | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 1 | 5 | 1 | 13
  Asian: Other | 1 | 0 | 1 | 0 | 5 | 0 | 2 | 0 | 0 | 0 | 0 | 9
  Asian: Unknown | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Asian: White | 26 | 15 | 24 | 13 | 26 | 10 | 30 | 31 | 10 | 26 | 10 | 221

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Clinical Response Measured by Simplified Hidradenitis Suppurativa (sHiSCR)
Description: sHiSCR was defined as at least a 50 percent (%) reduction in abscess and inflammatory nodule (AN) counts, and no increase in draining fistula count related to baseline. The primary variable was modeled with the binomial distribution. A neutral non-informative Beta (1/3, 1/3) distribution was used as the prior for the response rate for all treatment groups. Based on the priors and the observed primary outcome, posterior distributions for the response rate for the investigational treatment and pooled placebo groups were computed respectively. At the time of the statistical comparison for cohorts A, B, and C, the placebo data for cohorts D and E were incomplete and therefore excluded. Similarly, during the comparison for cohort D, the placebo data for cohort E was still pending and was not included.
Time Frame: Baseline, Week 16
Population: The Pharmacodynamic (PD) analysis set included all participants who received any study drug and had no protocol deviations with relevant impact on PD data.
Measure: Count of Participants; unit: Participants
Groups:
- Pooled Placebo (Cohorts A, B and C): Placebo to CFZ533, LYS006 and MAS825.
- Pooled Placebo (Cohorts A, B, C and D): Placebo to CFZ533, LYS006, MAS825 and LOU064.
- Pooled Placebo (Cohorts A, B, C, D and E): Placebo to CFZ533, LYS006, MAS825, LOU064 and VAY736.
Arm/Group | Cohort A - CFZ533 600 mg | Cohort B - LYS006 20 mg | Cohort C - MAS825 300 mg | Pooled Placebo (Cohorts A, B and C) | Cohort D - LOU064 25 mg | Cohort D - LOU064 100 mg | Pooled Placebo (Cohorts A, B, C and D) | Cohort E - VAY736 300 mg | Pooled Placebo (Cohorts A, B, C, D and E)
Number analyzed (Participants) | 29 | 25 | 32 | 39 | 33 | 33 | 49 | 31 | 60
Participants | 17 | 8 | 15 | 14 | 24 | 16 | 17 | 16 | 23
Statistical Analysis 1: Comparison: Cohort A - CFZ533 600 mg vs Pooled Placebo (Cohorts A, B and C); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Average difference in response rates = 22.1, 90% CI 2-sided [2.5 to 41.0] — 90% credible intervals of the treatment difference are reported as 90% Confidence Interval 2-Sided below
Statistical Analysis 2: Comparison: Cohort A - CFZ533 600 mg vs Pooled Placebo (Cohorts A, B and C); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Probability (%) diff. in resp. rate >= 0 = 97.1
Statistical Analysis 3: Comparison: Cohort B - LYS006 20 mg vs Pooled Placebo (Cohorts A, B and C); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Average difference in response rates = -3.3, 90% CI 2-sided [-21.9 to 15.9] — 90% credible intervals of the treatment difference are reported as 90% Confidence Interval 2-Sided below
Statistical Analysis 4: Comparison: Cohort B - LYS006 20 mg vs Pooled Placebo (Cohorts A, B and C); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Probability (%) diff. in resp. rate >= 0 = 38.7
Statistical Analysis 5: Comparison: Cohort C - MAS825 300 mg vs Pooled Placebo (Cohorts A, B and C); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Average difference in response rates = 12.2, 90% CI 2-sided [-7.5 to 31.6] — 90% credible intervals of the treatment difference are reported as 90% Confidence Interval 2-Sided below
Statistical Analysis 6: Comparison: Cohort C - MAS825 300 mg vs Pooled Placebo (Cohorts A, B and C); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Probability (%) diff. in resp. rate >= 0 = 84.7
Statistical Analysis 7: Comparison: Cohort D - LOU064 25 mg vs Pooled Placebo (Cohorts A, B, C and D); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Average difference in response rates = 37.2, 90% CI 2-sided [19.7 to 53.0] — 90% credible intervals of the treatment difference are reported as 90% Confidence Interval 2-Sided below
Statistical Analysis 8: Comparison: Cohort D - LOU064 25 mg vs Pooled Placebo (Cohorts A, B, C and D); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Probability (%) diff. in resp. rate >= 0 = 99.9
Statistical Analysis 9: Comparison: Cohort D - LOU064 100 mg vs Pooled Placebo (Cohorts A, B, C and D); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Average difference in response rates = 13.9, 90% CI 2-sided [-4.2 to 31.9] — 90% credible intervals of the treatment difference are reported as 90% Confidence Interval 2-Sided below
Statistical Analysis 10: Comparison: Cohort D - LOU064 100 mg vs Pooled Placebo (Cohorts A, B, C and D); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Probability (%) diff. in resp. rate >= 0 = 89.6
Statistical Analysis 11: Comparison: Cohort E - VAY736 300 mg vs Pooled Placebo (Cohorts A, B, C, D and E); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Average difference in response rates = 13.4, 90% CI 2-sided [-4.2 to 31.5] — 90% credible intervals of the treatment difference are reported as 90% Confidence Interval 2-Sided below
Statistical Analysis 12: Comparison: Cohort E - VAY736 300 mg vs Pooled Placebo (Cohorts A, B, C, D and E); Test type: Other — Bayesian Analysis using a Beta-binomial model; Bayesian Analysis; Probability (%) diff. in resp. rate >= 0 = 89.0

ADVERSE EVENTS:
Time Frame: Cohorts A, B and C: 28 weeks including 12 weeks follow up period. Cohort D: 20 weeks including 4 weeks follow up period. Cohort E (ongoing): up to 116 weeks including 100 weeks follow up period.
Groups:
- Total: Total
Arm/Group | Cohort A - CFZ533 600 mg | Cohort B - LYS006 20 mg | Cohort C - MAS825 300 mg | Cohort D - LOU064 25 mg | Cohort D - LOU064 100 mg | Cohort E - VAY736 300 mg | Pooled Placebo (Cohorts A, B, C, D and E) | Total
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27 | 0/33 | 0/33 | 0/33 | 0/32 | 0/61 | 0/248
Serious Adverse Events (participants affected / at risk) | 4/29 | 2/27 | 1/33 | 1/33 | 1/33 | 1/32 | 1/61 | 11/248
Other Adverse Events (participants affected / at risk) | 23/29 | 19/27 | 22/33 | 26/33 | 15/33 | 18/32 | 38/61 | 161/248
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - CFZ533 600 mg (N=29) | Cohort B - LYS006 20 mg (N=27) | Cohort C - MAS825 300 mg (N=33) | Cohort D - LOU064 25 mg (N=33) | Cohort D - LOU064 100 mg (N=33) | Cohort E - VAY736 300 mg (N=32) | Pooled Placebo (Cohorts A, B, C, D and E) (N=61) | Total (N=248)
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Abscess limb (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Genital abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Testicular torsion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A - CFZ533 600 mg (N=29) | Cohort B - LYS006 20 mg (N=27) | Cohort C - MAS825 300 mg (N=33) | Cohort D - LOU064 25 mg (N=33) | Cohort D - LOU064 100 mg (N=33) | Cohort E - VAY736 300 mg (N=32) | Pooled Placebo (Cohorts A, B, C, D and E) (N=61) | Total (N=248)
Increased tendency to bruise (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0 | 2 | 6
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 3 | 0 | 5 | 14
Flatulence (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 6
Asthenia (General disorders) | 3 | 0 | 2 | 2 | 0 | 0 | 4 | 11
Fatigue (General disorders) | 1 | 4 | 3 | 3 | 1 | 0 | 4 | 16
Pyrexia (General disorders) | 1 | 3 | 1 | 2 | 0 | 1 | 4 | 12
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 1 | 4
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 3 | 1 | 5
COVID-19 (Infections and infestations) | 3 | 1 | 8 | 2 | 2 | 0 | 3 | 19
Ear infection (Infections and infestations) | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 4
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 4 | 5
Nasopharyngitis (Infections and infestations) | 1 | 4 | 3 | 7 | 2 | 4 | 3 | 24
Sinusitis (Infections and infestations) | 2 | 0 | 3 | 0 | 0 | 1 | 1 | 7
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 6
Injection related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 6
Bacterial test positive (Investigations) | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 4
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 3
Blood glucose increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2
Blood urine present (Investigations) | 2 | 0 | 1 | 2 | 0 | 0 | 1 | 6
C-reactive protein increased (Investigations) | 0 | 0 | 2 | 2 | 0 | 0 | 3 | 7
Crystal urine present (Investigations) | 0 | 1 | 0 | 0 | 1 | 0 | 5 | 7
Nitrite urine present (Investigations) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Urine albumin/creatinine ratio increased (Investigations) | 2 | 3 | 1 | 1 | 1 | 0 | 2 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 1 | 0 | 0 | 2 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 0 | 0 | 0 | 1 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1 | 0 | 0 | 1 | 6
Dizziness (Nervous system disorders) | 1 | 2 | 0 | 2 | 1 | 0 | 1 | 7
Headache (Nervous system disorders) | 2 | 4 | 5 | 4 | 0 | 1 | 6 | 22
Depression (Psychiatric disorders) | 0 | 1 | 2 | 0 | 0 | 1 | 0 | 4
Proteinuria (Renal and urinary disorders) | 1 | 1 | 0 | 2 | 0 | 0 | 2 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 2 | 1 | 0 | 0 | 7
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 4
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 5 | 1 | 0 | 6 | 8 | 22
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 2 | 1 | 1 | 3 | 8
Hypertension (Vascular disorders) | 1 | 1 | 1 | 2 | 0 | 1 | 4 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2024-05-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT03827798/Prot_000.pdf
  • Statistical Analysis Plan (2025-02-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT03827798/SAP_001.pdf